CLINICAL TRIAL: NCT00014326
Title: A Phase III Randomized Study On Low-Dose Total Body Irradiation And Involved Field Radiotherapy In Patients With Localized, Stages I and II, Low Grade Non-Hodgkin's Lymphoma
Brief Title: Involved-Field Radiation Therapy in Treating Patients With Previously Untreated Stage I or Stage II Low-Grade Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-20971-22997; EORTC-20971; EORTC-22997
Record Dates: First submitted 2001-04-10; First posted 2003-01-27 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Lymphoma
Keywords: stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; contiguous stage II small lymphocytic lymphoma; contiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; nodal marginal zone B-cell lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Radiotherapy

INTERVENTIONS:
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Giving radiation therapy in different ways may kill more tumor cells. It is not yet known which regimen of radiation therapy is more effective for non-Hodgkin's lymphoma.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy to the involved area with or without total-body irradiation in treating patients who have low-grade stage I or stage II non-Hodgkin's lymphoma that has not previously been treated.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine if the addition of low-dose total body irradiation (TBI) to involved-field radiotherapy improves the disease-free survival of patients with previously untreated, stage I or II low-grade non-Hodgkin's lymphoma.
* Determine the response of patients treated with low-dose TBI.
* Compare the overall survival and quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, stage (I vs II), performance status (0-1 vs 2), lactate dehydrogenase elevation (yes vs no), histological subtype (small lymphocytic lymphoma vs lymphoplasmacytoid lymphoma vs follicular lymphoma), and, for stage I patients, presence of measurable mass (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo involved-field radiotherapy daily five days a week for 2.5-4 weeks.
* Arm II: Patients undergo low-dose total body irradiation (TBI) daily 5 days a week on weeks 1 and 4. At 4 weeks after completion of TBI, patients undergo involved-field radiotherapy as in arm I.

Quality of life is assessed before treatment, at 4 weeks after completion of involved-field radiotherapy, every 6 months for 5 years, and then annually thereafter.

Patients are followed every 3 months for 3 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 344 patients will be accrued for this study within 6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage I or II, low-grade, non-Hodgkin's lymphoma

  * Follicular lymphoma grade I, II, or III
  * Small lymphocytic lymphoma
  * Lymphoplasmacytoid lymphoma
  * Nodal marginal zone lymphoma
* Previously untreated disease
* At least 1 measurable or evaluable mass at least 1.1 cm (except for patients with stage I disease where the entire mass was removed for diagnostic purposes) NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 2,000/mm ^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other prior or concurrent malignancy except basal cell skin cancer or carcinoma in situ of the cervix
* No psychological, familial, sociological, or geographical condition that would preclude study participation
* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2001-01; Primary Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Disease-free survival

SECONDARY OUTCOMES:
Overall survival
Quality of life as assessed by European Organization of Research for the Treatment of Cancer (EORTC) Quality of Life Questionnaire (QoLQ) C30
Response as assessed by Cheson criteria

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Richaud, MD, Study Chair — Institut Bergonié; Marten Beijert, MD, Study Chair — University Medical Center Groningen, Groningen
Locations (15):
- Belgium (2):
  - U.Z. Gasthuisberg, Leuven
  - Universitair Medisch Centrum St. Radboud - Nijmegen, Leuven
- University Hospital Rebro, Zagreb, Croatia
- Rigshospitalet - Copenhagen University Hospital, Copenhagen, Denmark
- National Cancer Institute of Egypt, Cairo, Egypt
- France (5):
  - Centre D'Oncologie Du Pays-Basque, Bayonne
  - Institut Bergonie, Bordeaux
  - Centre Hospitalier de Dax, Dax
  - Hopital Robert Boulin, Libourne
  - Polyclinique Francheville, Périgueux
- Netherlands (5):
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - Maastro Clinic - Locatie Maastricht, Maastricht
  - Daniel Den Hoed Cancer Center at Erasmus Medical Center, Rotterdam
  - Dr. Bernard Verbeeten Instituut, Tilburg